CLINICAL TRIAL: NCT04917081
Title: 'Go With the Flow': Effects of Mindful Self-Compassion in Psychiatric Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: pro mente REHA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUGrazXXX
Record Dates: First submitted 2021-05-27; First posted 2021-06-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Meditation; Progressive Muscle Relaxation
Keywords: Mindful Self-Compassion
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Self-Compassion (Experimental)
  Interventions: Behavioral: Mindful Self-Compassion
- Progressive Muscle Relaxation (Active Comparator)
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Mindful Self-Compassion — Mindful Self-Compassion has been developed by Neff and Germer as a specific kind of Mindfulness-Based Interventions to promote self-compassion. It combines the skills of mindfulness and self-compassion, providing a powerful tool for emotional resilience and enhancing the capacity for emotional wellbeing. In this study, a shortened version of the MSC program is used which is applied once a week for 75 minutes throughout the patients' stay in the rehabilitation clinic.
  Arms: Mindful Self-Compassion
Behavioral: Progressive Muscle Relaxation — Progressive Muscle Relaxation by Jacobson is a deep relaxation technique that helps relieve muscle tension and is based on the premise that mental calmness is a natural result of physical relaxation. In this study, Progressive Muscle Relaxation is applied once a week for 75 minutes throughout the patients' stay in the rehabilitation clinic.
  Arms: Progressive Muscle Relaxation

SUMMARY:
This study is designed as a randomized controlled trial to gain further insights into possible effects of a standardized 6-week Mindful Self-Compassion (MSC) training on psychiatric rehabilitation inpatients and aims

* to generate insights into which parameters of mental health, and especially emotion regulation, can be improved by MSC in this setting,
* to compare effects of MSC training with an established relaxation training (i.e., progressive muscle relaxation; PMR) and
* to determine the general conditions and patient characteristics influencing the effectiveness of MSC training.

ELIGIBILITY:
Inclusion Criteria:

1. Psychiatric diagnosis
2. Signed informed consent form
3. Full command of the German language

Exclusion Criteria:

1. Age <18 years
2. Acute psychotic episode, acute suicidal tendencies, and acute addiction disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2021-08-11 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Change in Emotion Regulation Questionnaire (ERQ) | Baseline and 1 day after the last intervention
  The Emotion Regulation Questionnaire (ERQ) measures two common emotion regulation strategies (cognitive reappraisal and expressive suppression) with a total of 10 items (reappraisal scale: 6 items; suppression scale: 4 items), which are answered on a seven-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). The higher the score of a scale (mean value ranging from 1 to 7), the more frequently the respective emotion regulation strategy is used.
Change in Positive and Negative Affect Schedule (PANAS) | Baseline and 1 day after the last intervention
  The Positive and Negative Affect Schedule (PANAS) consists of 20 items and captures two dispositional dimensions (positive affect and negative affect), 10 items for each scale. A five-point Likert scale (1 - very slightly to 5 - extremely) is used. Mean scores for each of the two scales can range from 1 to 5, with lower scores representing lower levels of positive/negative affect and higher scores representing higher levels of positive/negative affect.
Reappraisal Inventiveness Test (RIT) | 1 day after the last intervention
  The Reappraisal Inventiveness Test (RIT) assesses emotion regulation abilities on a behavioral level. Participants generate cognitive reappraisals for different anger-provoking situations to reduce their anger. The fluency (total number of generated nonidentical ideas that qualified as cognitive reappraisals) and flexibility (number of categorically different reappraisals) of these reappraisals are measured. The given answers will be independently rated by two researchers. In addition, the intensity of induced anger will be assessed with a seven-point Likert scale from 0 (not at all) to 6 (very).

SECONDARY OUTCOMES:
Change in Self-Compassion Scale (SCS) | Baseline and 1 day after the last intervention
  SCS captures the amount of self-compassion by means of 26 items answered on a five-point Likert scale (1 to 5). A higher value (mean value ranging from 1 to 5) indicates a higher level of self-compassion.
Change in Short-Form-Health Survey (SF-12) | Baseline and 1 day after the last intervention
  SF-12 measures quality of life via 12 items answered with different response formats. The items are weighted and summed to provide a physical and mental health score ranging from 0 to 100, with a higher score indicating better health.
Change in Brief Symptom Inventory (BSI-18) | Baseline and 1 day after the last intervention
  The BSI-18 assesses psychiatric symptoms in three dimensions (somatization, depression and anxiety), which can be summarized in a global severity index (GSI). It contains 18 items that are answered on a five-point Likert scale ranging from 0 (not at all) to 4 (extremely). Higher values (ranging from 0 to 24 in the three dimensions; ranging from 0 to 72 in the GSI) indicate a greater severity of symptoms.
Change in Multidimensional Inventory for Religious/Spiritual Well-Being 12 (MI-RSB 12) | Baseline and 1 day after the last intervention
  The MI-RSB 12 captures four different dimensions of religious and spiritual well-being, namely general religiosity, forgiveness, connectedness, and immanent hope, which can be collated into a total amount of religious/spiritual well-being (RSB). The instrument consists of 12 items, three items per dimension, answered via a six-point Likert scale (1 - strongly disagree to 6 - strongly agree). Scores range from 3 to 18 for each subscale and from 12 to 72 for the overall score of the RSB. Higher scores indicate higher religious and spiritual well-being.
Change in Happiness | every day during the stay at the rehabilitation clinic
  The amount of subjective happiness will be captured by one item, which has to be answered on a 10-point Likert scale, with 1 indicating "not happy at all" and 10 "absolutely happy".

OTHER OUTCOMES:
Inventory of Personality Organization (IPO-16) | Baseline and 1 day after the last intervention
  Personality structure will be assessed with the IPO-16 which consists of the three subscales identity diffusion, primitive defenses, and reality testing. The 16 items (identity diffusion: 6 items; primitive defenses: 5 items; reality testing: 5 items) are rated on a five-point Likert scale ranging from 1 (never) to 5 (always). A global index is used for statistical analysis, which is gathered by the mean of all items and ranges between 1 and 5. A higher value indicates a higher structural impairment.
Experience in Close Relationships (Revised, German Version; ECR-RD12) | Baseline and 1 day after the last intervention
  To assess general attachment patterns, the ECR-RD12 will be used. This questionnaire assesses attachment-related anxiety (6 items) and attachment-related avoidance (6 items) with a total of 12 items, rated on a seven-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). Scale-scores range between 1 and 7. Higher scores on one or both dimensions are considered to indicate an insecure adult attachment orientation. Lower scores indicate a secure adult attachment orientation.
Sex | Baseline and 1 day after the last intervention
  Two questions are used to assess sex at birth and current sex with the following response options: 1 - female, 2 - male, 3 - transgender, 4 - other.
Age | Baseline
  Digit entry
Weight and Height (BMI) | Baseline and 1 day after the last intervention
  Weight (kg) and height (cm) will be assessed by digits entry and subsequently transformed into BMI.
Education | Baseline
  Education will be assessed via six response options (1 - compulsory education, 2 - completed apprenticeship, 3 - vocational high school, 4 - high school, 5 - college degree, 6 - university degree).
Employment | Baseline
  Employment will be assessed via four response options (1 - standing in the profession, 2 - in education, 3 - retired, 4 - without gainful employment).
Marital status | Baseline
  Marital status will be assessed via four response options (1 - married, 2 - partnership, 3 - single, 4 - widowed/divorced).
Confession | Baseline
  Confession will be assessed via six response options (1 - Christianity, 2 - Buddhism, 3 - Hinduism, 4 - Islam, 5 - none, 6 - other).
Children | Baseline
  Participants are asked whether they have children using a dichotomous response format (0 - no, 1- yes).
Diet | Baseline and 1 day after the last intervention
  Dietary habits will be assessed with the following response options: 1 - with a lot of meat, 2 - with little meat, 3 - with meat and rich in fruits and vegetables, 4 - vegetarian with fish and/or milk/eggs, 5 - vegan.
  In addition, it is also asked whether this diet has been followed for at least 6 months (0 - no, 1 - yes).
Cigarettes per day | Baseline and 1 day after the last intervention
  Digit entry
Alcohol consumption | Baseline and 1 day after the last intervention
  dichotomous response format (0 - no, 1 - yes)
Consumption of illegal drugs | Baseline and 1 day after the last intervention
  dichotomous response format (0 - no, 1 - yes)
Medication | Baseline and 1 day after the last intervention
  Medication will be assessed by free answer.
Mental illness | Baseline and 1 day after the last intervention
  Mental illness will be assessed by free answer.
Subjective feeling of health | Baseline and 1 day after the last intervention
  Subjective feeling of health will be captured via a ten-point rating scale (1 - not at all to 10 - absolutely).
Religiosity | Baseline and 1 day after the last intervention
  Religiosity will be captured via a ten-point rating scale (1 - not at all to 10 - absolutely).
Spirituality | Baseline and 1 day after the last intervention
  Spirituality will be captured via a ten-point rating scale (1 - not at all to 10 - absolutely).
Previous experience with meditation | Baseline
  dichotomous response format (0 - no, 1 - yes)
Previous experience with yoga | Baseline
  dichotomous response format (0 - no, 1 - yes)
Previous experience with mindfulness | Baseline
  dichotomous response format (0 - no, 1 - yes)
Previous experience with Progressive Muscle Relaxation (PMR) | Baseline
  dichotomous response format (0 - no, 1 - yes)
Previous experience with Mindful Self-Compassion (MSC) | Baseline
  dichotomous response format (0 - no, 1 - yes)
Practice of the learned practice (either PMR or MSC) | 1 day after the last intervention
  dichotomous response format (0 - no, 1 - yes); if answered with "yes" (I practice PMR/MSC) it is asked for the frequency of practice (1 - daily, 2 - several times a week, 3 - once a week, 4 - less than once a week), the duration of practice (1 - less than 10 minutes, 2 - 10-15 minutes, 3 - more than 15 minutes), and the type of practice (1 - ritualized, 2 - informal)
Sympathy of the learned practice (either PMR or MSC) | 1 day after the last intervention
  Subjective sympathy of the learned practice will be captured via a ten-point rating scale (1 - not at all to 10 - absolutely).
Sympathy of the trainer (either PMR or MSC) | 1 day after the last intervention
  Subjective sympathy of the trainer will be captured via a ten-point rating scale (1 - not at all to 10 - absolutely).

CONTACTS AND LOCATIONS:
Overall Officials: Human-Friedrich Unterrainer, PD DDr., Principal Investigator — Medical University Graz, Department of Psychiatry and Psychotherapeutic Medicine
Locations (1):
- pro mente REHA, Sonnenpark Neusiedlersee, Rust, Burgenland, Austria

IPD SHARING:
Plan to Share IPD: No